CLINICAL TRIAL: NCT06441825
Title: Patient Observation With Environmental and Wearable Sensors in Myasthenia Gravis
Acronym: POWER-MG
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Marc Günter Pawlitzki, Senior Physician, Heinrich-Heine University, Duesseldorf
Other Study IDs: MPGv1.0
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Myasthenia Gravis; Myasthenic Syndrome; Lambert-Eaton Myasthenic Syndrome
MeSH Terms: conditions — Myasthenia Gravis; Lambert-Eaton Myasthenic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — - Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myasthenic Syndromes Observational Cohort: Cohort to be characterized via clinical, serological and digital observations
  Interventions: Other: Increased multimodal observation including digital monitoring

INTERVENTIONS:
Other: Increased multimodal observation including digital monitoring — Digital monitoring combined with repeated clinical assessments and retrospective analysis of serological markers
  Other Names: Withings Scanwatch 2

SUMMARY:
This observational study seeks to investigate the underlying processes of myasthenia gravis by employing multimodal monitoring techniques. By integrating digital biomarkers alongside clinical monitoring, we aim to enhance the detection of disease activity and establish correlations between digital measures, clinical scores and various questionnaires including sores on quality of life, sleep quality or activities of daily living. Primarily including patients treated with newly approved drugs, it aims at improving and monitoring the efficacy and safety of treatment and allowing a more individualized treatment.

DETAILED DESCRIPTION:
Myasthenia Gravis (MG) is a chronic autoimmune disease characterized by muscle weakness and fatigue due to defective transmission at the neuromuscular junction. Typically, symptomatic assessments occur during clinical encounters, either as part of routine treatment assessments or in acute situations such as myasthenic crises. However, for a comprehensive understanding of mechanisms in MG and disease activity, continuous monitoring is essential.

Utilization of digital biomarkers derived from wearable devices offers unprecedented insights into diseases like MG and allows us to establish correlations between digital measures, clinical scores such as the QMG scale and MGC, as well as various questionnaires addressing sleep quality, quality of life or activities of daily living.

Data recorded by the used wearables (Withings Scanwatch 2) cover various parameters including activity-related data (step count, minutes in certain intensity levels), basic cardiovascular measurements such as heart rate, and sleep-related data (total time asleep, sleep quality, etc.).

Prospectively, this study aims at improving patient care by gaining a deeper insight into Myasthenia Gravis and its dynamic disease activity while concurrently monitoring the efficacy and safety of treatments, particularly of the newly approved drugs for MG.

In the future, wearables might hold the potential to improve treatment processes and optimize therapeutic approaches. For instance, digital biomarkers could serve as early warning signs for phenomena like heightened disease activity or end-of-dose phenomena, paving the way for personalized treatment strategies tailored to individual patient needs.

ELIGIBILITY:
* Formal diagnosis of generalized Myasthenia Gravis, with at least one of the following criteria:

  * Response to oral or intravenous administration of an acetylcholinesterase inhibitor
  * Evidence of pathological decrement/ elevated jitter
  * Evidence of Myasthenia Gravis-typical antibody (AChR, LRP4, MuSK, Titin) OR other diagnosed Myasthenic Syndrome
* Age ≥ 18
* Usage of Smartphone with Android 8.1 (or higher) or IOS12.3 (or higher)
* Able to provide informed consent, based on investigator´s judgment

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation:

* Unable or unwilling to give informed consent
* Unable or unwilling to use the smartphone app
* Any significant comorbidity that might potentially interfere with the ability to successfully participate in the study, based on investigator´s judgment
* Patient with exclusively ocular symptoms (ocular myasthenia gravis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myasthenic syndromes treated at the University Clinic Duesseldorf.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
QMG: Quantitative Myasthenia Gravis Scale | 6 months, monthly
  The QMG-Score is a clinical tool to assess the severity of symptoms in MG. It evaluates muscle strength and function in specific muscle groups (ocular, oral, facial, neck and limb muscles), grip strength and vital capacity. It ranges from 0 to 39, with higher scores indicating an increased symptom load.
MGC: Myasthenia Gravis Composite | Baseline, after 3 and 6 months
  The MGC is a clinical tool to evaluate the severity and progression of MG. It ranges from 0 to 50, with higher scores indicating a higher severity of MG.
MGFA-PIS: Myasthenia Gravis Post intervention status | Baseline, after 3 and 6 months
  The MGFA-PIS is a scoring system used to assess the status of patients with MG. It divides MG presentations into different classes, classifying outcome measures and treatment effectiveness. It has 8 classes; Minimal Manifestation can be further described within four dimensions.
MG-ADL: Myasthenia Gravis Activities of Daily Living | Baseline, after 3 and 6 months
  The MG-ADL is a tool used to assess the functional status of patients with MG in their daily activities. It consists of questions related to various activities of daily living such as speaking, chewing, swallowing, walking etc. It ranges from 0 to 24, with higher scores indicating a greater impairment in daily life.
MG-QoL15: Myasthenia Gravis Quality of Life-15 | Baseline, after 3 and 6 months
  The MG-QoL assesses the quality of life in patients with MG, covering various aspects of daily life such as physical functioning, social interactions, emotional well-being and overall satisfaction with life.
  It ranges from 0 to 60, with higher scores indicating a greater impact of MG on life quality.

SECONDARY OUTCOMES:
WHOQoL-BREF: World Health Organization Quality of Life Questionnaire Brief Version | Baseline, after 3 and 6 months
  The WHOQOL-BREF questionnaire measures quality of life across 4 domains: Physical health, psychological health, social relationships and environment. It also includes one question on overall QOL and one on general health. The WHOQOL-BREF scores correlate highly (.89 or above) with WHOQOL-100 scores, and demonstrate good discriminant validity, content validity, internal consistency and test-retest reliability. The four WHOQOL-BREF domain scores will be used as main outcome measure. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, with higher scores corresponding to greater QOL.
HADSD: Hospital Anxiety and Depression Scale | Baseline, after 3 and 6 months
  The HADSD is a self-assessment questionnaire measuring levels of anxiety and depression in patients. It contains two subscales: one for anxiety and one for depression. Total scores range from 0 to 42, with higher scores indicatiBAng higher levels of anxiety or depression.
EoD-Questionnaire: End of Dose-Questionnaire | Baseline, after 3 and 6 months
  The EoD-Questionnaire assesses the effectiveness of a treatment at the end of its dosing interval and asks about an increase in symptoms.
Sleep-Questionnaire: | Baseline, after 3 and 6 months
  The Sleep-Questionnaire contain the Pittsburgh Sleep Quality Index (PSQI) as well as two Items on the perceived impact of the smartwatch on the patient´s sleep. The PSQI assesses the quality of sleep over a one-month interval and measures seven component scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total score ranges from 0 to 21, with higher scores indicating a poorer sleep quality.
10. Questionnaire on Smartwatch Usage (after 6 Months) containing the System Usability Scale | After 6 months
Digital Measurements: Activity parameters - Longitudinal development of step count | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of approximate distance travelled (meter) | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of duration of soft activity (seconds) as defined by Withings | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of duration of moderate activity (seconds) as defined by Withings | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of duration of itnense activity (seconds) as defined by Withings | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of active time (seconds) as defined by Withings | 6 months, continuously
Digital Measurements: Activity parameters - longitudinal development of approximate calories burned as defined by Withings | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of time awake (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of number of times user woke up | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of time to sleep (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of total time asleep (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of total time in bed (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of ratio of sleep/time in bed | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of time spent in bed before falling asleep (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of time awake after first falling asleep (seconds) | 6 months, continuously
Digital Measurements: Sleep parameters - longitudinal development of Withings sleep Score as defined by Withings | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of average heartrate (beats/min) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of maximal heartrate (beats/min) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of minimum heartrate (beats/min) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of time in light heartrate zone (seconds) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of time in moderate heartrate zone (seconds) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of time in intense heartrate zone (seconds) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of time in maximal heartrate zone (seconds) | 6 months, continuously
Digital Measurements: Cardiovascular parameters - longitudinal development of heart rate variability (milliseconds) | 6 months, continuously
Smartwatch adherence | Continously 6 motnhs
  Wearing time of smartwatch (daily)

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine University, Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided